CLINICAL TRIAL: NCT00800488
Title: Usefulness of Serum Procalcitonin for Predicting Serious Bacterial Infection in Febrile Infants Less Than 3 Months
Brief Title: Procalcitonin for Predicting Serious Bacterial Infection in Infants Less Than 3 Months
Acronym: PRONOUR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 06 047
Record Dates: First submitted 2008-11-24; First posted 2008-12-02 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2011-04

CONDITIONS: Fever; Bacterial Infection
Keywords: Fever; Infant; Procalcitonin; Serious Bacterial Infection
MeSH Terms: conditions — Fever; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to study the value of serum procalcitonin as a predictive marker for severe bacterial infection in febrile infants.

2200 febrile infants aged less than 3 months will prospectively be included. All infants will have a measure of Procalcitonin concentrations. Comparison of the mean value of Procalcitonin concentration in infants with and without serious Bacterial infection.

Evaluation of the area under the ROC for Procalcitonin concentration.

DETAILED DESCRIPTION:
Serious bacterial infections are often difficult to detect in infant with fever without source. Procalcitonin is a better blood marker of infection than White blood cell count and possibly than C-reactive protein. This could lead to a reduction in antibiotic prescription. Our objective is to evaluate the impact of Procalcitonin result on antibiotic prescription in children 1 to 3 month old with fever without source and our hypothesis is that it will lower the antibiotic prescription rate.

ELIGIBILITY:
Inclusion Criteria:

* Infant older than 7 days old and less than 3 months old.
* Fever (defined by a rectal temperature greater than or equal to 38°C)
* Emergency consultation

Exclusion Criteria:

* Infants with a previously identified immunodeficiency or chronic disease,
* Antibiotic treatment within the previous 48 hours

Ages: 7 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 7 days older to 3 month older with fever
Sampling Method: Non-Probability Sample
Enrollment: 2209 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve of the serum Procalcitonin concentration in the diagnosis of serious bacterial infections | At the day of emergency consultation for fever

SECONDARY OUTCOMES:
Diagnostic value (sensibility and specificity) of clinical examination versus procalcitonin | At the day of emergency consultation for fever
Diagnostic value (sensibility and specificity) of complete blood count versus procalcitonin | At the day of emergency consultation for fever
Diagnostic value (sensibility and specificity) of CRP versus procalcitonin | At the day of emergency consultation for fever

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAJDOS, MD, Principal Investigator — Assistance Publique-Hôpitaux de Paris, Hôpital Antoine Béclère
Locations (1):
- Pediatric Emergency Depatment - Hôpital Antoine Béclère, Clamart, Hauts-de-Seine, France